CLINICAL TRIAL: NCT05627544
Title: Blood Transfusion Applications in Hip Replacements: A Retrospective Study
Brief Title: Blood Transfusion Applications in Hip Replacements
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yonca Özvardar Pekcan, MD, Anesthesia and Reanimation specialist, principal investigator, Baskent University
Other Study IDs: KA22/430
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Blood Transfusion; Hip Replacement; Anesthesia Management
Keywords: Blood Transfusion; Hip Replacement; Anesthesia
MeSH Terms: interventions — Demography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First 6 year group: Patients who underwent hip replacement between 2010 and 2016 by the same experienced surgeon in our hospital
  Interventions: Procedure: Anesthesia management/Hip replacement surgery; Procedure: Demographic data; Procedure: Chronic diseases; Procedure: Postoperative complication
- Second 6 year group: Patients who underwent hip replacement between 2017 and 2022 by the same experienced surgeon in our hospital
  Interventions: Procedure: Anesthesia management/Hip replacement surgery; Procedure: Demographic data; Procedure: Chronic diseases; Procedure: Postoperative complication

INTERVENTIONS:
Procedure: Anesthesia management/Hip replacement surgery — The effect of anesthesia management on blood transfusion practices in hip replacement surgeries
Procedure: Demographic data — The effect of demographic data on blood transfusion practices in hip replacement surgeries
Procedure: Chronic diseases — The effect of chronic diseases on blood transfusion practices in hip replacement surgeries
Procedure: Postoperative complication — The effect of blood transfusion applications on postoperative complications in hip replacement surgeries

SUMMARY:
Introduction and Aim In the intraoperative or postoperative period of hip replacement surgeries, approximately 46% of patients receive erythrocyte transfusion. 'Patient blood management' protocols have been established in order to reduce the frequency of perioperative surgical bleeding and transfusion. The aim of this study is to evaluate the patients who underwent hip replacement by the same experienced surgeon; to evaluate retrospectively in terms of patient characteristics, surgical and anesthesia management, blood transfusion frequency.

Methods The characteristics of patients who underwent hip replacement (total hip replacement, revision hip replacement, partial hip replacement) operation by the same experienced surgeon between 2010-2022 at Baskent University after the approval of Baskent University Medical and Health Sciences Research Board, results will be analyzed retrospectively through perioperative follow-up forms and review of patient files.

Expectations and scientific contributions Preparing patients for surgery, determining the causes of blood loss during and after surgery and creating preventive strategies are important for all operations, especially hip replacement surgeries. While determining the strategies, the main aim should be to see the pre-, intra- and post-operative period as a whole, to determine the transfusion risks according to the comorbidities and anemia of the patients, and to determine the anesthesia and analgesia managements that reduce blood loss in the intraoperative and postoperative periods.

DETAILED DESCRIPTION:
Introduction and Aim Hip replacement surgeries are among the operations whose frequency is increasing in our country and in the world. In these operations, procedures such as soft tissue dissection, exposing the hypervascular metaphysis and bone resection cause acute blood loss and continue in the form of leakage in the postoperative period. It has been reported that the rate of blood transfusion in hip operations in the United States is between 18-68%. There are studies reporting that erythrocyte transfusion rate approximately 46% of these cases in the intraoperative or postoperative period. Various complications may develop in patients during or after blood transfusion. These complications include local or systemic infections, venous thromboembolic events, allergic reactions, circulatory overload, transfusion-induced acute lung injury, morbidity, mortality, and increased hospital stay. In addition, a significant increase in cost can be seen. It is thought that the amount of bleeding varies according to the duration of the operation, the experience of the surgeon, and the type of surgery. Therefore, it is important for patient safety to reduce surgical bleeding and avoid transfusion applications as much as possible.

"Patient blood management" has been defined as, to reduce the frequency of perioperative surgical bleeding and transfusion. Perioperative patient blood management practices, correction of preoperative anemia, autologous blood donation, discontinuation of blood thinners, acute normovolemic hemodilution, use of tranexamic acid, regional anesthesia, controlled hypotension, avoidance of hypothermia, appropriate fluid management, meticulous surgery, appropriate hemostasis, patient position, postoperative drain strategy. 'Patient blood management' measures are actively applied in hip replacement surgeries, which are one of the major orthopedic surgeries.

The aim of this study is to evaluate the patients who underwent hip replacement by the same experienced surgeon in this center; to evaluate retrospectively in terms of patient characteristics, surgical and anesthesia management, blood transfusion frequency.

Methods The characteristics of patients who underwent hip replacement (total hip replacement, revision hip replacement, partial hip replacement) operation by the same experienced surgeon between 2010-2022 at Baskent University after the approval of Baskent University Medical and Health Sciences Research Board, It will be analyzed retrospectively through perioperative follow-up forms and review of patient files.

From preoperative records; Demographic data (Age, sex, height, body weight), diagnoses (Hip arthrosis, hip revision, hip fracture, congenital hip dislocation, infected hip replacement revision), American Society of Anesthesiologists Physical Condition Classification (ASA), co-morbidities (Hypertension, diabetes, chronic kidney failure, hepatopathy, inflammatory disease), smoking, alcohol, antiplatelet/anticoagulant, nonsteroidal anti-inflammatory use (NSAII), opioid, herbal medicine use, antiplatelet cut-off time compliance, hemoglobin (Hb), hematocrit (Htc), leukocytes, thrombocyte, activated partial thromboplastin time (APTT), prothrombin time (PTZ), international normalized ratio (INR), preoperative erythrocyte (ES) transfusion/amount.

From intraoperative records; Year of operation, mallampati score, type of operation, duration of operation, whether emergency or elective, duration of anesthesia, type of anesthesia, intraoperative blood pressure (systolic and diastolic), heart rate, peripheral oxygen saturation, amount/type of fluid administered, ES transfusion/ amount, Hb when transfused, drugs used for anesthesia and analgesia and their amount, amount of blood in the aspirator, administration of tranexamic acid, amount of intraoperative urine.

From the postoperative records; Hb/Htc values, ES transfusion/amount/day of administration, use of drain, amount of blood in the drain, amount of postoperative urine, intensive care unit admission, initiation of anticoagulants, early and late complications (Atrial fibrillation, pneumonia , renal failure, prosthesis infection, allergic reactions, nausea-vomiting), postoperative analgesia (Epidural/intravenous patient-controlled analgesia, opioid and NSAID use), Hb, urea, creatinine values at postoperative 6th and 12th hours and at discharge, iron preparation use, The number of hospitalization days and the mortality within 7 days will be recorded and the data will be compared.

Statistical analysis Statistical analysis will be performed using SPSS (SPSS Inc. Chicago, Illinois, USA) version 20.0 of the statistical program. Descriptive statistical methods (frequency, percentage, mean, standard deviation) will be used while evaluating the study data. The Kolmogorov-Smirnov test will be used to evaluate the conformity of the data of the patients with and without ES transfusion to normal distribution. T-test will be used in the analysis of data suitable for normal distribution, Kruskal-Wallis test or Mann Whitney U test will be used in the analysis of data not suitable for normal distribution. X² will be used in the analysis of qualitative or counted data. p<0.05 will be considered significant.

Expectations and scientific contributions Preparing patients for surgery, determining the causes of blood loss during and after surgery and creating preventive strategies are important for all operations, especially hip replacement surgeries. While determining the strategies, the main aim should be to see the pre-, intra- and post-operative period as a whole, to determine the transfusion risks according to the comorbidities and anemia of the patients, and to determine the anesthesia and analgesia managements that reduce blood loss in the intraoperative and postoperative periods. With this study, it is aimed to both update the practice and contribute to the literature by examining the operations performed by the same experienced surgeon and testing the effectiveness and safety of the strategies applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone hip replacement by the same experienced surgeon in the last 12 years

Exclusion Criteria:

* Patients with insufficient data will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone hip replacement by the same experienced surgeon in the last 12 years will be retrospectively screened from patient files and the system in terms of anesthesia and blood transfusion applications.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Amount of preoperative, peroperative and postoperative blood transfusion | Up to 1 week
  The amount of blood transfusion administered to patients who have undergone hip replacement surgery by the same experienced surgeon in the last 12 years will be measured and compared during their hospitalization.

SECONDARY OUTCOMES:
Anesthesia management | Up to 1 week
  The effects of preoperative preparation for surgery, anesthesia applications during the operation, and analgesia applications in the postoperative period on the amount of blood transfusion in patients hospitalized for hip replacement surgery will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca Özvardar Pekcan, Principal Investigator — Baskent University
Locations (1):
- Baskent University Zubeyde Hanim Practice and Research Center, Izmir, Karşıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen AB, Mehnert F, Overgaard S, Johnsen SP. Allogeneic blood transfusion and prognosis following total hip replacement: a population-based follow up study. BMC Musculoskelet Disord. 2009 Dec 29;10:167. doi: 10.1186/1471-2474-10-167. PMID 20040083
- [Background] Browne JA, Adib F, Brown TE, Novicoff WM. Transfusion rates are increasing following total hip arthroplasty: risk factors and outcomes. J Arthroplasty. 2013 Sep;28(8 Suppl):34-7. doi: 10.1016/j.arth.2013.03.035. Epub 2013 Jul 26. PMID 23896359
- [Background] Ponnusamy KE, Kim TJ, Khanuja HS. Perioperative blood transfusions in orthopaedic surgery. J Bone Joint Surg Am. 2014 Nov 5;96(21):1836-44. doi: 10.2106/JBJS.N.00128. PMID 25378512
- [Background] Song K, Pan P, Yao Y, Jiang T, Jiang Q. The incidence and risk factors for allogenic blood transfusion in total knee and hip arthroplasty. J Orthop Surg Res. 2019 Aug 28;14(1):273. doi: 10.1186/s13018-019-1329-0. PMID 31455380
- [Background] Menendez ME, Lu N, Huybrechts KF, Ring D, Barnes CL, Ladha K, Bateman BT. Variation in Use of Blood Transfusion in Primary Total Hip and Knee Arthroplasties. J Arthroplasty. 2016 Dec;31(12):2757-2763.e2. doi: 10.1016/j.arth.2016.05.022. Epub 2016 May 18. PMID 27325367
- [Background] Carling MS, Jeppsson A, Eriksson BI, Brisby H. Transfusions and blood loss in total hip and knee arthroplasty: a prospective observational study. J Orthop Surg Res. 2015 Mar 28;10:48. doi: 10.1186/s13018-015-0188-6. PMID 25889413
- [Background] Saleh A, Small T, Chandran Pillai AL, Schiltz NK, Klika AK, Barsoum WK. Allogenic blood transfusion following total hip arthroplasty: results from the nationwide inpatient sample, 2000 to 2009. J Bone Joint Surg Am. 2014 Sep 17;96(18):e155. doi: 10.2106/JBJS.M.00825. PMID 25232085
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Taylor RW, Manganaro L, O'Brien J, Trottier SJ, Parkar N, Veremakis C. Impact of allogenic packed red blood cell transfusion on nosocomial infection rates in the critically ill patient. Crit Care Med. 2002 Oct;30(10):2249-54. doi: 10.1097/00003246-200210000-00012. PMID 12394952
- [Background] Tezcan B. Etkin hasta kan yönetimi. JARSS 2019; 27: 162-73.
- [Background] Spahn DR. Anemia and patient blood management in hip and knee surgery: a systematic review of the literature. Anesthesiology. 2010 Aug;113(2):482-95. doi: 10.1097/ALN.0b013e3181e08e97. PMID 20613475
- [Background] Artroplasty Society of Australia. Guidelines for venous thrombotic episode prophylaxis for hip and knee arthroplasty. Australian Orthopaedic Association 2010
- [Background] Tuttle JR, Ritterman SA, Cassidy DB, Anazonwu WA, Froehlich JA, Rubin LE. Cost benefit analysis of topical tranexamic acid in primary total hip and knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1512-5. doi: 10.1016/j.arth.2014.01.031. Epub 2014 Feb 3. PMID 24630599